CLINICAL TRIAL: NCT02802735
Title: A Phase 1, Open-label, Two Part Study to Evaluate the Pharmacokinetics of Single and Multiple Doses of Apremilast in Healthy Adult Male Korean Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of Single and Multiple Doses of Apremilast in Healthy Adult Male Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-CP-033
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics; Apremilast; Healthy Adult Male; Korean Subjects
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Part 1 of the study was a 3-treatment period, 3-sequence crossover study. Part 2 was a parallel-group, placebo-controlled, single-period study.
Masking Description: Part 1 was a randomized open-label crossover study. Part 2 was a randomized, double-blind study.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: Apremilast 20 mg (Experimental): A single oral dose of 20 mg apremilast.
  Interventions: Drug: Apremilast
- Part 1: Apremilast 30 mg (Experimental): A single oral dose of 30 mg apremilast.
  Interventions: Drug: Apremilast
- Part 1: Apremilast 40 mg (Experimental): A single oral dose of 40 mg apremilast.
  Interventions: Drug: Apremilast
- Part 2: Apremilast 30 mg BID (Experimental): 30 mg apremilast orally twice a day (BID) for 14 days.
  Interventions: Drug: Apremilast
- Part 2: Placebo (Placebo Comparator): Matching placebo orally twice a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Tablet for oral administration
  Other Names: CC-10004; OTEZLA®
  Arms: Part 1: Apremilast 20 mg; Part 1: Apremilast 30 mg; Part 1: Apremilast 40 mg; Part 2: Apremilast 30 mg BID
Drug: Placebo — Tablet for oral administration
  Arms: Part 2: Placebo

SUMMARY:
This two-part study was designed to evaluate the pharmacokinetics (PK) of single and multiple doses of apremilast in healthy adult Korean males.

DETAILED DESCRIPTION:
The study will consist of two parts. Part 1 will evaluate the PK of ascending single doses of apremilast. Part 2 will evaluate the PK of apremilast when administered as multiple doses over 14 days.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must satisfy the following criteria to be enrolled in the study:

1. Healthy adult male Korean subjects between 18 and 45 years of age (inclusive) at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Must be able to communicate with the Investigator and understand and comply with the requirements of the study.
5. Must be in good health as determined by the Investigator according to past medical history, physical examination (PE), vital signs, 12-lead electrocardiogram (ECG), and laboratory tests.
6. Must have a body mass index (BMI) between 18 and 30 kg/m^2 (inclusive).
7. Clinical laboratory tests must be within normal limits or considered by the Investigator to be not clinically significant.
8. Vital signs (systolic and diastolic blood pressure, pulse rate, and oral [or tympanic] body temperature) will be assessed in the supine position after the subject has rested for at least five minutes. Subject must be afebrile (febrile [oral or tympanic] is defined as ≥ 38°C or 100.3°F) with vital signs within the following ranges:

   * Systolic blood pressure: 90 to 140 mm Hg;
   * Diastolic blood pressure: 50 to 90 mm Hg;
   * Pulse rate: 40 to 110 bpm.
9. Must have a normal or clinically acceptable 12-lead ECG. Subjects must have a QTc value ≤ 450 msec.
10. Must have a normal or clinically acceptable physical examination.
11. Contraception Requirements:

    - Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex or non-latex condoms NOT made out of natural [animal] membrane [for example, polyurethane]) while on Investigational Product (IP) and for at least 28 days after the last dose of investigational product (IP).
12. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study, and for at least 28 days after the last dose of IP.

Exclusion Criteria:

* The presence of any of the following will exclude any healthy subject from enrollment into the study:

  1. History of any clinically significant and relevant neurological, psychiatric, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.
  2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
  3. Use of any prescribed systemic or topical medication within 30 days of the first dose administration.
  4. Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.
  5. Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, colon resection, irritable bowel syndrome, Crohn's disease, etc. Subjects with cholecystectomy and appendectomy may be included.
  6. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
  7. Donated blood or plasma within eight weeks before the first dose administration to a blood bank or blood donation center.
  8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs.
  9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or a positive alcohol screen.
  10. Known to have hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies, or have a positive result to the test for HBsAg, HCV antibodies or human immunodeficiency virus (HIV) antibodies at Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT02802735?term=CC-10004-CP-033&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-part study in healthy Korean men. The study was conducted at 1 clinic in Korea.
Pre-assignment Details: In Part 1 participants were randomized to 1 of 3 treatment sequences consisting of 3 treatment periods.
  In Part 2 participants were randomized in a 3:1 ratio to receive apremilast or matching placebo twice a day (BID) for 14 days.
Groups:
- Part 1: Apremilast 20 mg / 30 mg / 40 mg: Participants received a single oral dose of 20 mg apremilast on day 1 of period 1, a single oral dose of 30 mg apremilast on day 1 of period 2, and a single oral dose of 40 mg apremilast on day 1 of period 3. There was a 7-10 day washout period between each dose.
- Part 1: Apremilast 30 mg / 20 mg / 40 mg: Participants received a single oral dose of 30 mg apremilast on day 1 of period 1, a single oral dose of 20 mg apremilast on day 1 of period 2, and a single oral dose of 40 mg apremilast on day 1 of period 3. There was a 7-10 day washout period between each dose.
- Part 1: Apremilast 40 mg / 20 mg / 30 mg: Participants received a single oral dose of 40 mg apremilast on day 1 of period 1, a single oral dose of 20 mg apremilast on day 1 of period 2, and a single oral dose of 30 mg apremilast on day 1 of period 3. There was a 7-10 day washout period between each dose.
- Part 2: Apremilast 30 mg BID: Participants received 30 mg apremilast orally twice a day for 14 days.
- Part 2: Placebo BID: Participants received matching placebo orally twice a day for 14 days.
Period: Overall Study
Arm/Group | Part 1: Apremilast 20 mg / 30 mg / 40 mg | Part 1: Apremilast 30 mg / 20 mg / 40 mg | Part 1: Apremilast 40 mg / 20 mg / 30 mg | Part 2: Apremilast 30 mg BID | Part 2: Placebo BID
Started | 4 | 4 | 4 | 12 | 4
Completed | 4 | 3 | 4 | 12 | 4
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Part 1: Apremilast: Participants received a single oral dose of 20 mg apremilast, 30 mg apremilast, and 40 mg apremilast across 3 treatment periods separated by a washout period of 7-10 days.
- Total: Total of all reporting groups
Arm/Group | Part 1: Apremilast | Part 2: Apremilast 30 mg BID | Part 2: Placebo BID | Total
Number analyzed (Participants) | 12 | 12 | 4 | 28
Age, Continuous [Mean (Full Range); unit: years] | 29.8 [19.0 to 43.0] | 30.8 [24.0 to 41.0] | 25.5 [20.0 to 31.0] | 29.6 [19.0 to 43.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 12 | 4 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 12 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: Concentrations of apremilast in plasma were measured using a validated liquid chromatography tandem mass spectrometry assay.
Time Frame: Day 1 of each treatment period at predose (0 hour) and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60, and 72 hours post-dose.
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1: Apremilast 20 mg: Participants received a single oral dose of 20 mg apremilast.
- Part 1: Apremilast 30 mg: Participants received a single oral dose of 30 mg apremilast.
- Part 1: Apremilast 40 mg: Participants received a single oral dose of 40 mg apremilast.
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
ng/mL | 205 (32.1) | 273 (32.1) | 373 (19.7)

2. Primary Outcome: Part 1: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
hours | 3.0 [1.5 to 5.0] | 3.0 [1.5 to 5.0] | 2.0 [0.5 to 5.0]

3. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) for Apremilast
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
ng*hr/mL | 1770 (25.8) | 2330 (22.6) | 3470 (25.7)

4. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) for Apremilast
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
ng*hr/mL | 1790 (25.5) | 2360 (22.1) | 3500 (25.6)

5. Primary Outcome: Part 1: Terminal Elimination Half-life (T1/2) for Apremilast
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
hours | 7.4 (35.2) | 8.2 (44.4) | 7.4 (36.8)

6. Primary Outcome: Part 1: Apparent Clearance of Apremilast From Plasma After Extravascular Administration (CL/F)
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
liters/hour | 11.1 (25.5) | 12.7 (22.1) | 11.4 (25.6)

7. Primary Outcome: Part 1: Apparent Volume of Distribution of Apremilast During the Terminal Phase (Vz/F)
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg
Number analyzed (Participants) | 11 | 12 | 12
liters | 120 (47.6) | 151 (49.6) | 122 (38.7)

8. Primary Outcome: Part 2: Area Under the Plasma Concentration-time Curve During a Dosage Interval (AUCτ) for Apremilast
Description: Area under the plasma concentration-time curve during a dosage interval (tau) at steady state, where tau is 12 hours.
Time Frame: Day 1 and day 14 prior to the morning dose (0 hour), and at 0.5, 1, 1.5, 2, 3, 5, 8, and 12 hours after the morning dose
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 2: Apremilast 30 mg BID: Participants received 30 mg apremilast orally twice a day (BID) for 14 days.
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
ng*hr/mL
  Day 1 | 1610 (33.0)
  Day 14 | 2600 (34.3)

9. Primary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Time Frame: as for outcome 8
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
ng/mL
  Day 1 | 283 (34.3)
  Day 14 | 408 (36.5)

10. Primary Outcome: Part 2: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Time Frame: as for outcome 8
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
hours
  Day 1 | 2.00 [1.00 to 5.00]
  Day 14 | 1.50 [1.00 to 3.00]

11. Primary Outcome: Part 2: Terminal Elimination Half-life (T1/2) for Apremilast
Time Frame: Day 14 prior to the morning dose (0 hour), and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60, and 72 hours after the morning dose
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
hours | 7.80 (31.4)

12. Primary Outcome: Part 2: Apparent Clearance of Apremilast From Plasma After Extravascular Administration (CL/F)
Time Frame: as for outcome 11
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
liters/hour | 11.5 (34.3)

13. Primary Outcome: Part 2: Apparent Volume of Distribution of Apremilast During the Terminal Phase (Vz/F)
Time Frame: as for outcome 11
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
liters | 130 (53.3)

14. Primary Outcome: Part 2: Ratio of Accumulation
Description: Ratio of accumulation calculated as Day 14 AUC0-τ / Day 1 AUC0-τ
Time Frame: Day 1 and day 14 prior to the morning dose (0 hour), and at 0.5, 1, 1.5, 2, 3, 5, 8, and 12 hours after the morning dose, and on day 14 only at 24, 36, 48, 60, and 72 hours after the morning dose
Population: Participants who received at least 1 dose of apremilast and had at least 1 measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 2: Apremilast 30 mg BID
Number analyzed (Participants) | 12
ratio | 1.62 (36.0)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Time Frame: Part 1, up to 40 days; Part 2, up to 24 days
Population: Participants who received at least 1 dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg | Part 2: Apremilast 30 mg BID | Part 2: Placebo BID
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 4
Participants
  Any treatment-emergent adverse event (TEAE) | 2 | 1 | 3 | 7 | 3
  TEAE related to study drug | 1 | 1 | 2 | 6 | 2
  Serious adverse events | 0 | 0 | 0 | 0 | 0
  Serious adverse events related o study dug | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation | 0 | 0 | 0 | 0 | 0
  Treatment-related TEAE leading to discontinuation | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1, up to 40 days; Part 2, up to 24 days
Groups:
- Part 1: Total: Participants received a single oral dose of 20 mg apremilast, 30 mg apremilast, and 40 mg apremilast across 3 treatment periods separated by a washout period of 7-10 days.
- Part 2: Total: Participants who received 30 mg apremilast or placebo twice a day for 14 days
Arm/Group | Part 1: Apremilast 20 mg | Part 1: Apremilast 30 mg | Part 1: Apremilast 40 mg | Part 1: Total | Part 2: Apremilast 30 mg BID | Part 2: Placebo BID | Part 2: Total
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/12 | 0/12 | 0/4 | 0/16
Other Adverse Events (participants affected / at risk) | 2/11 | 1/12 | 3/12 | 4/12 | 7/12 | 3/4 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Apremilast 20 mg (N=11) | Part 1: Apremilast 30 mg (N=12) | Part 1: Apremilast 40 mg (N=12) | Part 1: Total (N=12) | Part 2: Apremilast 30 mg BID (N=12) | Part 2: Placebo BID (N=4) | Part 2: Total (N=16)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 4
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.